CLINICAL TRIAL: NCT00260351
Title: Immunogenicity and Safety of Purified Vero Cell Rabies Vaccine (PVRV, Verorab™) Administered for Rabies Post-exposure Treatment. Comparison of Essen-IM, Zagreb-IM, and Thai Red Cross (TRC)-ID Regimens in the Indian Population.
Brief Title: Immunogenicity and Safety of Verorab™ in Indian Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAB28
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Rabies
Keywords: rabies;; rabies post-exposure;; category III
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Participants on Thai Red Cross, TRC-ID regimen
  Interventions: Biological: Purified Verocell Rabies Vaccine
- Group 2 (Experimental): Participants on Zagreb-IM regimen
  Interventions: Biological: Purified Verocell Rabies Vaccine
- Group 3 (Experimental): Participants on Essen-IM regimen.
  Interventions: Biological: Purified Verocell Rabies Vaccine

INTERVENTIONS:
Biological: Purified Verocell Rabies Vaccine — 0.1 mL, ID (TRC regimen)
  Other Names: PVRV, VERORAB
  Arms: Group 1
Biological: Purified Verocell Rabies Vaccine — 0.5 mL, IM (ZAGREB regimen)
  Other Names: PVRV, VERORAB
  Arms: Group 2
Biological: Purified Verocell Rabies Vaccine — 0.5 mL, IM (ESSEN regimen)
  Other Names: PVRV, VERORAB
  Arms: Group 3

SUMMARY:
* To demonstrate that rabies vaccine administered according to the Thai Red Cross, (TRC)-ID regimen (2-2-2-0-1-1) is not inferior to rabies vaccine administered according to the ESSEN IM regimen in terms of Geometric Mean Titers (GMTs) at D28, in subjects with a WHO category III rabies exposure,or,
* To demonstrate that Rabies vaccine administered according to the ZAGREB-IM regimen (2-1-1) is not inferior to Rabies vaccine administered according to the ESSEN IM regimen in terms of GMTs at D28, in subjects with a WHO category III rabies exposure.

Secondary objectives:

1. To describe the immunogenicity profile of each regimen
2. To assess the safety of the vaccine in each group.

ELIGIBILITY:
Inclusion Criteria:

* Subject with WHO category III rabies exposure
* Subject aged at least 2 years old (day of second birthday)

Exclusion Criteria:

* Subject unable to comply with the follow-up schedule of the protocol
* Delayed post-exposure treatment (>72 hours between incident and treatment
* Subject bitten by an observable animal at the inclusion visit
* Subject with immune-compromised or underlying diseases which may lead to inferior immune response
* Subject with known pregnancy at the time of inclusion
* Subject enrolled or scheduled to be enrolled in another clinical study.
* Subject with acute febrile illness/ axillary temperature > 37.5 degree celsius
* Subject in whom blood sampling will be difficult.
* Subject receiving chloroquine or other anti-malarial treatment
* Subject receiving immunosuppressive therapy, other immune-modifying drug or cytotoxic drugs
* Subject with known chronic illnesses (ie. heart, lung, kidney, liver) including immunosuppressive diseases (cancer, HIV, etc.)
* Previous rabies immunization
* Subject having received any vaccine within the previous 30 days, except tetanus toxoid and tetanus immunoglobulin
* Subject with clinical signs of rabies
* Subject with known allergy to vaccine components (e.g. neomycin)
* Subject who received blood and/or plasma transfusion within the past 3 months

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2004-12; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: To provide information concerning the immune response of Purified Verocell Rabies Vaccine | 6 months post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (3):
- India (3):
  - Hyderabad
  - Kolkata
  - Lucknow

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com